CLINICAL TRIAL: NCT03609073
Title: A Prospective Study to Evaluate the Safety and Feasibility of an Endoluminal-suturing Device (Endomina TM) as an Aid for Diverticulum Treatment
Brief Title: Endomina Diverticulum
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: enrollment too slow
Sponsor: Erasme University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P2018/262
Record Dates: First submitted 2018-06-11; First posted 2018-08-01 (Actual); Last update posted 2021-11-24 (Actual); Status verified 2021-11

CONDITIONS: Oesophageal Disease
Keywords: endoscopy; mini invasive
MeSH Terms: conditions — Esophageal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental)
  Interventions: Device: Endomina

INTERVENTIONS:
Device: Endomina — Suturing system then cutting the bridge between the diverticulum and the esophagus.

SUMMARY:
Esophageal diverticulum is a rare disease. Majority comes form the pharyngo-esophageal junction (70 % Zenker's Diverticulum), 10% are mediothoracic and 20% epiphrenic. Zenker's diverticulum is well treated with endoscopy (efficacy around 80%, complications around 5%) (1). For medio or epihrenic diverticulum, the classic treatment is surgery (diverticulectomy with or without anti-reflux surgery) but is associated with 33% morbidity and 9% mortality (2). Recently another technique involving magnet was described (3). Five patients were treated with success.

Considering the surgical risk, other techniques need to be evaluated. Using the Endomina device, sutures can be apposed between the foot of the diverticulum and the esophageal lumen. If necessary the bridge between the diverticulum and the esophagus can be cut with needle knife as described in Zenker's diverticulum treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Symptomatic medio or epiphrenic diverticulum.
2. Age between 18-80 years;
3. Must be able to comply with all study requirements for the duration of the study as outlined in the protocol. This includes complying with the visit schedule as well as study specific procedures such as: clinical assessment, endoscopy, radiography, as well as laboratory investigations;
4. Must be able to understand and be willing to provide written informed consent;
5. Must live within 75 km of the treatment site;

Exclusion Criteria:

1. Achalasia and any other esophageal motility disorders.
2. Severe esophagitis
3. Gastro-duodenal ulcer
4. Severe renal, hepatic, pulmonary disease or cancer;
5. GI stenosis or obstruction;
6. Pregnancy, breastfeeding or willing to become pregnant in the coming 18 months;
7. Anticoagulant therapy;
8. Currently participating in other study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2018-03-06 (Actual); Primary Completion 2021-10-25 (Actual); Study Completion 2021-10-25 (Actual)

PRIMARY OUTCOMES:
Incidence of all Adverse Device Effects | one year from procedure
  Safety will be characterized by the incidence of all Adverse Device Effects

SECONDARY OUTCOMES:
Dysphagia | one year from procedure
  Efficacy will be measured by the Dakkak and Bennett score of Dysphagia (Score 0 - no dysphagia to 4 - aphagia)

CONTACTS AND LOCATIONS:
Locations (1):
- Gastroenterology Department Erasme Hospital, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No